CLINICAL TRIAL: NCT05107570
Title: Cold-induced Thermogenesis in Adults From Siberia and Western Europe
Brief Title: The Effect of Cold Exposure on Energy Expenditure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: WEU
Record Dates: First submitted 2021-09-21; First posted 2021-11-04 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Cold Exposure
Keywords: Cold exposure; Energy expenditure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold exposure applied to Western European individuals (Other): Participants rested under thermoneutral conditions for 30 min, which was then followed by exposure to ~ 9°C air temperature for a maximum of 1 hour. Same duration as matched Siberian individuals.
  Interventions: Other: Cold exposure
- Cold exposure applied to Siberian individuals (Other): Participants rested under thermoneutral conditions for 30 min, which was then followed by exposure to ~ 9°C air temperature for a maximum of 1 hour. Same duration as matched European individuals.
  Interventions: Other: Cold exposure

INTERVENTIONS:
Other: Cold exposure — Cold air exposure (~ 9°C, maximum 1 hour duration)

SUMMARY:
Cold-induced thermogenesis, or the increase in energy expenditure upon cold exposure, indicates metabolic stress, as such, cold-induced thermogenesis may signal an appropriate stimulus to improve metabolic health. Cold acclimation may alter cold-induced thermogenesis due to changes in (non)shivering thermogenesis and blood flow. The main aim of this research is to compare the energy expenditure responses, during a standardised cold stress (~ 9°C air temperature, maximum 1 hour), of Siberian adults with Western European adults. The subjects will be individually matched for age, sex, body mass and height. It was hypothesised that cold-induced thermogenesis will be reduced in the Siberian population.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Western European origin or of Siberian origin
* BMI between 18.5 and 35 kg/m2
* Generally healthy (determined by dependent physician)

Exclusion Criteria:

* Smoking
* Active, uncontrolled cardiovascular disease or cancer
* Raynaud's disease
* Participation in another biomedical study within 1 month before the first study
* Cold-acclimated (Western European group), such as takes daily extended cold baths, works in a refrigerated environment, or regular cold-water swimming within 1 month of starting the study
* Medication use known to hamper subject's safety during study procedures
* Abuse of alcohol or drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
Cold-induced thermogenesis | 30 min before and during the cold exposure (maximum 1 hour)
  Energy expenditure with indirect calorimetry

SECONDARY OUTCOMES:
Skin temperature | 30 min before and during the cold exposure (maximum 1 hour)
  Skin temperature determined with iButtons, measured in °C
Core temperature | 30 min before and during the cold exposure (maximum 1 hour)
  Core temperature determined with a gastrointestinal pill, measured in °C
Shivering activity | 30 min before and during the cold exposure (maximum 1 hour)
  Electromyography will be used to measure the electrical activity of 3 skeletal muscles
Substrate oxidation | 30 min before and during the cold exposure (maximum 1 hour)
  Carbohydrate and fat oxidation will be determined with indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: W. van Marken Lichtenbelt, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Netherlands